CLINICAL TRIAL: NCT06042140
Title: Cryopreserved Human Umbilical Cord as a Meningeal Patch in Fetoscopic Spina Bifida Repair: Single Arm Phase III Trial.
Brief Title: Cryopreserved Human Umbilical Cord as a Meningeal Patch in Fetoscopic Spina Bifida Repair
Acronym: HUC-FICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ramesha Papanna, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0584; 1R01HD119340-01 (NIH)
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Spina Bifida; Fetus; Myelomeningocele; Myeloschisis
Keywords: Fetoscopic fetal intervention; Human umbilical cord; NEOX Cord 1K
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NEOX Cord 1K applied fetoscopically (Experimental): Patients intending to undergo open in-utero spina bifida repair will be offered to be screened for an alternative minimally invasive approach. All eligible pregnant mothers' fetuses within the trial will receive NEOX Cord 1K® as a spinal cord cover to close the developmental defect. In some cases, at the discretion of the Pediatric Neurosurgeon, NEOX Cord 1K® may be required to cover the skin. All eligible subjects meeting all inclusion criteria but none of the exclusion criteria may be enrolled.
  Interventions: Device: NEOX Cord 1K applied fetoscopically

INTERVENTIONS:
Device: NEOX Cord 1K applied fetoscopically — Under general anesthesia and tocolysis, in-utero repair begins with a laparotomy that is followed by exteriorization of the uterus. The fetus is then positioned by external cephalic version. Uterine entry will be accessed using 3 cannulas, followed by heated-humidified carbon dioxide insufflation for visualization. Then, fetoscopically the placode will be examined and dissected. The lesion will be repaired using NEOX Cord 1K® (HUC) for closure of the first layer over the neural placode. Primary closure of the skin will then occur, or NEOX Cord 1K® (human umbilical cord) will be used for skin closure at the discretion of the Pediatric Neurosurgeon. Finally, the laparotomy site will be sutured in multiple layers.

SUMMARY:
The objective is to test the efficacy of a laparotomy-assisted fetoscopic surgical approach to cover spina bifida spinal cord developmental defects using cryopreserved human umbilical cords (NEOX Cord 1K®) as a meningeal and skin patch.

ELIGIBILITY:
Inclusion Criteria:

Maternal Inclusion Criteria:

1. Singleton pregnancy
2. Gestational age at screening is 19 to 25 5/7 weeks and gestational age at surgery is 22 to 25 6/7 weeks
3. Maternal age: 18 years and older
4. Body mass index ≤45 kg/m2 (pre-pregnancy)
5. No preterm birth risk factors (short cervix <20 mm or a history of previous preterm delivery)
6. No previous uterine incision in the active uterine segment
7. Willing to undergo an open fetal repair if the fetoscopic approach is unsuccessful

Fetal Inclusion Criteria:

1. Spina bifida defect between T1 to S1 vertebral levels
2. Chiari II malformation
3. No evidence of kyphosis (curved spine)
4. No major life-threatening fetal anomaly unrelated to spina bifida
5. Normal karyotype, or a normal chromosomal microarray analysis (CMA), or a CMA with variants of unknown significance [fluorescence in situ hybridization (FISH) acceptable if ≥ 24 weeks].

Exclusion Criteria:

Maternal Exclusion Criteria:

1. Non-resident of the United States
2. Multifetal pregnancy
3. Poorly controlled insulin-dependent pregestational diabetes
4. Poorly controlled A2 diabetes mellitus (A2DM) insulin-dependent diabetes
5. Current or planned cerclage or documented history of an incompetent cervix
6. Placenta previa or placental abruption
7. Short cervix of < 20 mm
8. Obesity as defined by a body mass index of > 45 kg/m2
9. Previous spontaneous singleton delivery prior to 37 weeks
10. Maternal-fetal Rh isoimmunization, Kell sensitization, or a history of neonatal alloimmune thrombocytopenia
11. HIV or Hepatitis-B positive status
12. Known Hepatitis-C positivity
13. Uterine anomaly such as large or multiple fibroids or a mullerian duct abnormality that is diagnosed via imaging prior to surgery, which that are unavoidable during surgery
14. Other medical conditions which are contraindication to surgery or general anesthesia
15. Patient does not have a support person
16. Inability to comply with the travel and follow-up requirements of the trial
17. Patient does not meet psychosocial standardized assessment criteria
18. Participation in this or another intervention study that influences maternal and fetal morbidity and mortality
19. Maternal hypertension
20. Zika virus positivity
21. Allergy/history of drug reaction to Amphotericin B

Fetal exclusion criteria:

1. Major fetal anomaly not related to spina bifida
2. Kyphosis in the fetus of 30 degrees or more
3. Ventriculomegaly greater than 15 mm and no movements noted at hip and knee joints

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2031-03-08 (Estimated); Study Completion 2036-09-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants that can ambulate independently by walking at least 10 steps | 30-36 months after delivery

SECONDARY OUTCOMES:
Number of participants with lower extremity motor and sensory levels exceeding the anatomical level of the lesion by ≥ 2 segments | 30-36 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ramesha Papanna, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No